CLINICAL TRIAL: NCT05793762
Title: Evaluation of the Impact of Laterality on Cerebral Activation During a Virtual Mirror Therapy Task of Upper Limb Using fNIRS Technology in Healthy Subjects
Brief Title: Evaluation of the Impact of Laterality on Brain Activation During a Virtual Mirror Therapy Task in Healthy Subjects
Acronym: LARTHEMIRS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2022-17
Record Dates: First submitted 2023-03-08; First posted 2023-03-31 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: mirror therapy; laterality; cortical activation; functional near-infrared spectroscopy; upper limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: 30 right handed healthy participants aged between 18 and 60.
  Interventions: Device: Left virtual mirror therapy task; Device: Right virtual mirror therapy task

INTERVENTIONS:
Device: Left virtual mirror therapy task — the participant is seated on a chair facing the screen of the virtual mirror therapy device. both hands resting under the screen. The participant is asked, for each block of 20 seconds, to observe the visual feedback of the virtual left hand on the screen (flexion / extension movements of the fingers at 0.5 Hz).
Device: Right virtual mirror therapy task — the participant is seated on a chair facing the screen of the virtual mirror therapy device. both hands resting under the screen. The participant is asked, for each block of 20 seconds, to observe the visual feedback of the virtual right hand on the screen (flexion / extension movements of the fingers at 0.5 Hz).

SUMMARY:
The aim of this study is to investigate the differences in brain activation in healthy subjects during virtual mirror therapy tasks, depending on the laterality of the task. It seems that mirror therapy-related brain activation is greater when the visual feedback represents the non-dominant hand. The aim of this study is to highlight brain activation profiles during the use of virtual mirror therapy according to the lateralization of the feedback.

DETAILED DESCRIPTION:
Stroke frequently leads to upper limb deficit. The recovery of motor skills depends on many factors including laterality. The literature shows that cerebral activation during motor tasks differs depending on whether one is right-handed or left-handed and whether one uses the dominant hand or not. These differences probably lead to different recovery mechanisms depending on the side of the lesion and the laterality. An imaging technique is particularly suitable for exploring these different mechanisms: fNIRS (Functional Near Infra Red Spectroscopy). This method allows (like fMRI) to study cerebral neurovascular coupling. It is based on the fact that an activated brain region increases its local blood flow. Oxygenated (HbO) and deoxygenated (HbR) hemoglobin absorb infrared light and it is then possible to identify the cerebral cortical regions involved in a given task. This technique therefore makes it possible to study cerebral activation under more ecological conditions than fMRI and is thus particularly suitable for exploring rehabilitation techniques.

This research aims to study and compare in healthy subjects, using an fNIRS apparatus, the brain regions involved in a virtual mirror therapy task according to the laterality of the task.

The investigations will be carried out by the principal investigator or by specialized technicians from the neurology functional exploration department.

The acquisition has a duration of 15 minutes, it begins with a rest period of 120 seconds, which corresponds to the baseline. two different tasks are performed during the acquisition for each subject:

* observation of visual feedback of the right hand (RVF)
* observation of visual feedback of the left hand (LVF)

The design is a block design, each task, which has a duration of 20 seconds, is carried out 10 times per acquisition. There is therefore a total of 20 tasks whose order will be randomized.

Before each acquisition, the movements of the right and left hands (finger flexion and extension) are recorded by a camera integrated in the virtual mirror therapy tool. Movements are performed at a frequency of 0.5 Hz which appears to be the optimal frequency for observing cortical activation using a metronome.

Between periods of movement, the subject is in a rest position for a period from 15 to 25 seconds.

The instructions given to each subject are to observe the visual feedback on the screen and not to perform any movement during the acquisition.

After recruiting the subjects, the study investigator will check the inclusion and exclusion criteria.

If the subject can integrate the protocol, the acquisition will then be planned.

On the day of the acquisition, the fNIRS acquisition helmet (Brite MKII) will be installed by a specialist technician and instructions will be given. The recording is then made.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 60
* Right handed
* No neurological disease

Exclusion Criteria:

* Person under tutorship or curatorship
* Known allergy to components of the fNIRS device: neoprene

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: right handed healthy subjects aged between 18 and 60
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Mean change in the concentration of oxyhemoglobin during the task | Baseline
  Changes in the concentration of oxyhemoglobin during the task measured with fnirs device
Mean change in the concentration of deoxyhemoglobin during the task | Baseline
  Changes in the concentration of deoxyhemoglobin during the task measured with fnirs device

SECONDARY OUTCOMES:
Compare the cortical regions involved during the different mirror therapy tasks | Baseline
  visual analog scale.
Compare the feelings of the subjects | Baseline
  visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Julien BONNAL, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Bartur G, Pratt H, Dickstein R, Frenkel-Toledo S, Geva A, Soroker N. Electrophysiological manifestations of mirror visual feedback during manual movement. Brain Res. 2015 May 5;1606:113-24. doi: 10.1016/j.brainres.2015.02.029. Epub 2015 Feb 23. PMID 25721791
- [Background] Altschuler EL, Wisdom SB, Stone L, Foster C, Galasko D, Llewellyn DM, Ramachandran VS. Rehabilitation of hemiparesis after stroke with a mirror. Lancet. 1999 Jun 12;353(9169):2035-6. doi: 10.1016/s0140-6736(99)00920-4. No abstract available. PMID 10376620
- [Background] Chang CS, Lo YY, Chen CL, Lee HM, Chiang WC, Li PC. Alternative Motor Task-Based Pattern Training With a Digital Mirror Therapy System Enhances Sensorimotor Signal Rhythms Post-stroke. Front Neurol. 2019 Nov 22;10:1227. doi: 10.3389/fneur.2019.01227. eCollection 2019. PMID 31824406
- [Background] Ferrari M, Quaresima V. A brief review on the history of human functional near-infrared spectroscopy (fNIRS) development and fields of application. Neuroimage. 2012 Nov 1;63(2):921-35. doi: 10.1016/j.neuroimage.2012.03.049. Epub 2012 Mar 28. PMID 22510258
- [Background] Giraux P, Sirigu A. Illusory movements of the paralyzed limb restore motor cortex activity. Neuroimage. 2003 Nov;20 Suppl 1:S107-11. doi: 10.1016/j.neuroimage.2003.09.024. PMID 14597303
- [Background] Lee SH, Jin SH, An J. The difference in cortical activation pattern for complex motor skills: A functional near- infrared spectroscopy study. Sci Rep. 2019 Oct 1;9(1):14066. doi: 10.1038/s41598-019-50644-9. PMID 31575954
- [Background] Michielsen ME, Selles RW, van der Geest JN, Eckhardt M, Yavuzer G, Stam HJ, Smits M, Ribbers GM, Bussmann JB. Motor recovery and cortical reorganization after mirror therapy in chronic stroke patients: a phase II randomized controlled trial. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):223-33. doi: 10.1177/1545968310385127. Epub 2010 Nov 4. PMID 21051765
- [Background] Ramachandran VS, Rogers-Ramachandran D, Cobb S. Touching the phantom limb. Nature. 1995 Oct 12;377(6549):489-90. doi: 10.1038/377489a0. No abstract available. PMID 7566144
- [Background] Thieme H, Morkisch N, Mehrholz J, Pohl M, Behrens J, Borgetto B, Dohle C. Mirror therapy for improving motor function after stroke. Cochrane Database Syst Rev. 2018 Jul 11;7(7):CD008449. doi: 10.1002/14651858.CD008449.pub3. PMID 29993119
- [Background] Wang J, Fritzsch C, Bernarding J, Krause T, Mauritz KH, Brunetti M, Dohle C. Cerebral activation evoked by the mirror illusion of the hand in stroke patients compared to normal subjects. NeuroRehabilitation. 2013;33(4):593-603. doi: 10.3233/NRE-130999. PMID 24018372